CLINICAL TRIAL: NCT02137525
Title: A Randomized, Multicenter, Double-Blind, Double Dummy, Active Comparator, Dose-Ranging Study to Explore the Efficacy of SUBSYS® in Emergency Department Patients With Acute Pain
Brief Title: Study to Explore Effectiveness of Sublingual Fentanyl Spray in Emergency Department Patients With Acute Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was never initiated
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INS-14-022
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Morphine; Intravital Microscopy; Standard of Care; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Morphine 6 mg (Active Comparator): Placebo Sublingual Spray (PSS) + Intravenous Morphine (IVM 6 mg), every 30 minutes for two hours as needed (or until rescue), maximum exposure morphine 30 mg
  Interventions: Drug: Morphine 6 mg; Drug: Placebo Sublingual Spray
- Fentanyl 100 µg (Experimental): Intravenous Placebo (IVP) + Fentanyl Sublingual Spray (FSS 100 µg), every 30 minutes for two hours as needed (or until rescue), maximum exposure fentanyl 500 µg
  Interventions: Drug: Fentanyl 100 µg; Drug: Intravenous Placebo
- Fentanyl 200 µg (Experimental): Intravenous Placebo (IVP) + Fentanyl Sublingual Spray (FSS 200 µg), every 30 minutes for two hours as needed (or until rescue), maximum exposure fentanyl 1000 µg
  Interventions: Drug: Fentanyl 200 µg; Drug: Intravenous Placebo
- Fentanyl 400 µg (Experimental): Intravenous Placebo (IVP) + Fentanyl Sublingual Spray (FSS 400 µg), every 30 minutes for two hours as needed (or until rescue), maximum exposure fentanyl 2000 µg
  Interventions: Drug: Fentanyl 400 µg; Drug: Intravenous Placebo

INTERVENTIONS:
Drug: Morphine 6 mg — Intravenous infusion - delivering morphine 6 mg
  Other Names: IVM 6 mg; Standard of Care
  Arms: Morphine 6 mg
Drug: Fentanyl 100 µg — Fentanyl sublingual spray - single unit delivering 100 µg fentanyl
  Other Names: FSS 100 µg; SUBSYS®
  Arms: Fentanyl 100 µg
Drug: Fentanyl 200 µg — Fentanyl sublingual spray - single unit delivering 200 µg fentanyl
  Other Names: FSS 200 µg; SUBSYS®
  Arms: Fentanyl 200 µg
Drug: Fentanyl 400 µg — Fentanyl sublingual spray - single unit delivering 400 µg fentanyl
  Other Names: FSS 400 µg; SUBSYS®
  Arms: Fentanyl 400 µg
Drug: Placebo Sublingual Spray — Matching sublingual spray - single unit delivering 0 µg fentanyl
  Other Names: PSS
  Arms: Morphine 6 mg
Drug: Intravenous Placebo — Matching intravenous infusion - delivering 0 mg morphine
  Other Names: IVP
  Arms: Fentanyl 100 µg; Fentanyl 200 µg; Fentanyl 400 µg

SUMMARY:
This study will explore effectiveness of three doses of fentanyl sublingual spray against an active comparator in emergency department (ED) patients with acute pain.

After screening, eligible participants will participate in a treatment period (up to 2 hours) and a post-treatment evaluation period (up to 4 hours or discharge from the ED). Open-label standard of care rescue medication for pain can be given at any time during the study period, based on clinical judgment of the treating physician.

Adverse events will be collected for five days after initial enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Is able to understand the language in which the study is being conducted and has provided meaningful written informed consent for the study
* Has an acute painful condition requiring parenteral analgesia as deemed necessary by the treating physician or physician extender
* Has a pain score within protocol-specified parameters

Exclusion Criteria:

* Has allergy to fentanyl or morphine
* Has oxygen-dependent conditions or oxygen saturation <95%
* Has planned or recent drug use outside protocol-specified parameters
* Has any condition that, in the principal investigator's opinion, would place the patient at risk or influence the conduct of the study or interpretation of results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage of participants requiring additional doses of randomized pain medication | at 30 minutes after initial treatment

SECONDARY OUTCOMES:
Percentage of participants requiring additional doses of randomized pain medication at secondary time points | within 120 minutes after initial treatment
Visual analogue scale (VAS) Summed Pain Intensity Difference (SPID) calculated as Area under the Curve (AUC) every 30 minutes | from baseline through 120 minutes after the initial dose of investigational product
Number of Investigational Product (IP) administrations | within 120 minutes after initial treatment
Time to onset of pain relief (in minutes) using the stopwatch method | within 120 minutes after first treatment
Richmond Agitation Sedation Scale (RASS) score | within 120 minutes after first treatment
Percentage of Participants requiring rescue medication | during the 5-day study period
Time until rescue medication was required | during the 5-day study period
Percentage of participants experiencing a treatment-related adverse event | during the 5-day study period
Percentage of participants with clinically significant changes in vital signs | during the 5-day study period

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni DeCastro, Study Director — INSYS Therapeutics Inc
Locations (15):
- United States (15):
  - Maricopa Medical Center, Phoenix, Arizona
  - Olive View-UCLA Medical Center, Sylmar, California
  - Kansas University Medical Center, Kansas City, Kansas
  - Henry Ford Hospital, Detroit, Michigan
  - Wayne State University School of Medicine, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Stony Brook University HSC, Stony Brook, New York
  - Duke University School of Medicine, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia